CLINICAL TRIAL: NCT05267717
Title: Impact of Pessary Treatment on Cervical Stiffness Measurement and Birth Outcomes in Patients at Risk for Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asklepios proresearch (Industry)
Collaborators: AG Pregnolia (Unknown)
Responsible Party: Sponsor
Other Study IDs: #4011
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-01

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Cervical stiffness; Risk assessment; Pregnolia System
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control/Normal (no-pessary) group: All participants will must meet the criteria in order to be eligible: a singleton gestation, pregnant women recruited between 18+0 - 24+6 weeks of gestation, maternal age ≥18 years, the ability to sign approved consent form to participate in the study.
  Moreover for a normal cohort are being enrolled only asymptomatic pregnant women with no risk factors for spontaneous preterm birth
  Interventions: Other: Non-interventional study, all patients being tested with AG Pregnolia System to assess the values of the Cervical Stiffness
- Pessarry group: All participants will must meet the criteria in order to be eligible: a singleton gestation, pregnant women recruited between 18+0 - 24+6 weeks of gestation, maternal age ≥18 years, the ability to sign approved consent form to participate in the study.
  Moreover both for a pessary cohort additional cohort-specific criteria need to be met. Those are: suspected short cervix and confirmotian with transvaginal ultrasound - TVUS (CL < 3rd percentile at gestational age at measurement) according to Salomon at al.
  Interventions: Other: Non-interventional study, all patients being tested with AG Pregnolia System to assess the values of the Cervical Stiffness

INTERVENTIONS:
Other: Non-interventional study, all patients being tested with AG Pregnolia System to assess the values of the Cervical Stiffness — Non-interventional study,

SUMMARY:
Background: A preterm birth remain a worldwide important socioeconomic burden since prematurity has been consistently implicated in a wide range of health medical problems affecting newborn child and contributed in up to more than a half of overall perinatal mortality. Several studies have shown a significant therapeutic benefit as a result of an antenatal cervical pessary use in a high-risk preterm birth group of pregnant women. However the underlying mechanism by which pessary can reduce a risk of a preterm birth remain elusive. The study aims to quantitatively assess an ectocervical stiffness in a normal and in a treated with a pessary high-risk preterm birth pregnancy.

Methods: A prospective, non-interventional, post-market, monocentric, longitudinal, cohort study in a obstetric-led tertiary maternity teaching hospital to determine ectocervical stiffness and its changes measured prior and after the placement of a pessary, and the correlation of measured cervical stiffness or its changes with birth outcome in a high-risk preterm birth pregnant women indicated for cervical pessary. A cervical stiffness measured with Pregnolia system as the Cervical Stiffness Index (CSI, in mbar) will be a primary, whilst patient delivery data (gestational age, mode of delivery and complications) will be a secondary endpoint. In this pilot study, up to 142 subjects will be enrolled to have a total of 120 subjects (estimated dropout rate of 15%) completed the study; Pessary cohort: 60 (up to 71 recruited), normal cohort: 60 (up to 71 recruited).

Discussion: We hypothesize than the study will substantially improve our knowledge about cervical incontinency and preterm labour pathophysiology. We hope that our investigation will be able to elucidate ectocervical stiffness phenomenon both in high-risk preterm birth and in normal pregnant control, as well as the impact of cervical pessary use on a the CSI values.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the criteria in order to be eligible: a singleton gestation, pregnant women recruited between 18+0 - 24+6 weeks of gestation, maternal age ≥18 years, the ability to sign approved consent form to participate in the study.

Moreover both for a pessary cohort and for a normal cohort additional cohort-specific criteria for each group will need to be met. For the pessary cohort those shall consist of: suspected short cervix and confirmed on TVUS (CL < 3rd percentile at gestational age at measurement) according to Salomon at al, whilst for the control (no-pessary) group: asymptomatic pregnant women with no risk factors for spontaneous preterm birth, respectively

Exclusion Criteria:

Any possible exclusion criteria will be evaluated for an ineligibility for the study on a first visit. Exclusion criteria for both pessary and control group will be: evidence of fetal anomaly or fetal chromosomal abnormality from fetal ultrasound, uterine malformations, a history of diethylstilboestrol (DES) use, (cases of so-called so called DES daughters, who were exposed to DES in utero), a cervical cerclage or pessary currently in place, a silicone allergy, painful regular contractions, abnormal placentation (previa, accrete), the rupture of membranes, a cervical dilation, any visible, symptomatic cervical or vaginal infections (this excludes treated, asymptomatic infections), a known HIV infection, cervical carcinoma, the presence on the cervix at the 12 o'clock position of any of the following conditions: Nabothian cyst, cervical myomas, cervical condylomas, cervical endometriosis, cervical tears, scar tissue, cervical ectopy, cervical scarring due to prior LLETZ, cervical squamous intraepithelial lesion, cervical dysplasia, cone biopsy, a vaginal bleeding evident on exam.

The exclusion criteria about conditions on the cervix at 12 o'clock position cannot be checked without being enrolled in the study as it is an extra study assessment. Therefore, participants will be enrolled, the speculum assessment will be done after enrolment to clarify if any condition on the cervix at 12 o'clock position according to the exclusion criterion is present. If yes, the woman needs to be excluded from the study shortly after enrolment. These subjects will be replaced to reach the total number calculated.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only pregnant women
Study Population: Study population Determining a study eligibility will occur on a first visit. Since our research will be longitudinal and cohort study, two cohorts of subjects to enable a cross group differences comparison will be distinguished: the pessary and the normal (non-pessary) cohort.
  Sample size calculation In this pilot study, up to 142 subjects will be enrolled to have a total of 120 subjects (estimated dropout rate of 15%) completed the study; Pessary cohort: 60 (up to 71 recruited), normal cohort: 60 (up to 71 recruited). Currently, it is difficult to perform a formal power analysis since the primarx System is a novel device and limited underlying clinical data exists.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Stiffness Index | The first visit (18+0-24+6 weeks of gestation) and the follow-up visit (4 weeks later)
  The primary objective is to determine the absolute value of CSI (Cervical Stiffness Index) and its change over time in women undergoing pessary treatment, in comparison to normal pregnancies, when measured at 18+0 to 24+6 weeks and at the follow-up visit (4 weeks later).

SECONDARY OUTCOMES:
the correlation of the initial CSI and CSI changes with birth outcome | The first visit (18+0-24+6 weeks of gestation) and the follow-up visit (4 weeks later)
  The secondary objective is to determine the correlation of the initial CSI and CSI changes with birth outcome (gestational age at birth). The safety objective is the safety of the device, by assessing incidence, severity and seriousness of device-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- ASKLEPIOS proresearch, Department of Pre-and Perinatal Medicine, Asklepios Barmbek, Hamburg-Barmbek, Germany., Hamburg, Lohmühlenstraße 5/Haus J,, Germany

IPD SHARING:
Plan to Share IPD: Undecided